CLINICAL TRIAL: NCT01782352
Title: Age-related Macular Degeneration (AMD) in the Vitamin D and Omega-3 Trial (VITAL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, William G. Christen, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P001797; R01EY021900 (NIH); 2012P000724 (Other: Brigham and Women's Hospital)
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration; incidence; progression
MeSH Terms: conditions — Macular Degeneration; Disease Progression | interventions — Fatty Acids, Omega-3; Fish Oils; Omacor; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil placebo (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator): Vitamin D placebo
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3 placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Vitamin D placebo
  fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo
- Vitamin D + fish oil (Active Comparator): Vitamin D (cholecalciferol), 2000 IU per day
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Omega-3 fatty acids (fish oil)
  Other Names: Omacor
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Dietary Supplement: Vitamin D3 placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 Trial (VITAL; NCT 01169259) is a randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or omega-3 fatty acids, compared to placebo, reduce the incidence and/or progression of age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This ancillary study to the VITamin D and OmegA-3 TriaL (VITAL) will examine whether vitamin D3 and omega-3 fatty acids can help prevent the onset or progression of age-related macular degeneration (AMD). The study will also examine whether vitamin D3 and omega-3 fatty acids interact with each other, or with specific genes associated with AMD or vitamin D3 or omega-3 fatty acid metabolic activity, to affect the risk of developing AMD.

ELIGIBILITY:
Inclusion Criteria:

* All participants in VITAL (NCT 01169259) are eligible to participate in this ancillary study.

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2010-07; Primary Completion 2019-12 (Actual); Study Completion 2024-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Debra A Schaumberg, ScD, Principal Investigator — Brigham and Women's Hospital; William G Christen, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Christen WG, Cook NR, Manson JE, Buring JE, Chasman DI, Lee IM, Bubes V, Li C, Haubourg M, Schaumberg DA; VITAL Research Group. Effect of Vitamin D and omega-3 Fatty Acid Supplementation on Risk of Age-Related Macular Degeneration: An Ancillary Study of the VITAL Randomized Clinical Trial. JAMA Ophthalmol. 2020 Dec 1;138(12):1280-1289. doi: 10.1001/jamaophthalmol.2020.4409. PMID 33119047
- See also: VITAL study website — http://vitalstudy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 401605 initially screened; 39430 eligible to enter run-in; 25871 eligible for randomization; 2x2 factorial design: 12927 assigned to active vit D (of these, 6463 were assigned to active omega-3 FAs and 6464 to placebo omega-3 FAs) & 12944 assigned to placebo vit D (of these, 6470 were assigned to active omega-3 FAs and 6474 to placebo omega-3 FAs)
Pre-assignment Details: The trial included a 3-month placebo run-in period to select participants likely to have excellent compliance. Only individuals who reported taking at least 2/3 of their study pills during the run-in and met other eligibility criteria were randomized into the trial.
Groups:
- Vitamin D + Fish Oil: Vitamin D (cholecalciferol), 2000 IU per day
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Omega-3 fatty acids (fish oil)
  Vitamin D3
- Vitamin D + Fish Oil Placebo: Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo
  Vitamin D3
  Fish oil placebo
- Vitamin D Placebo + Fish Oil: Vitamin D placebo
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Omega-3 fatty acids (fish oil)
  Vitamin D3 placebo
- Vitamin D Placebo + Fish Oil Placebo: Vitamin D placebo
  fish oil placebo
  Vitamin D3 placebo
  Fish oil placebo
Period: Overall Study
Arm/Group | Vitamin D + Fish Oil | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo
Started | 6463 | 6464 | 6470 | 6474
Completed | 6463 | 6464 | 6470 | 6474
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Fish Oil | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Total
Number analyzed (Participants) | 6463 | 6464 | 6470 | 6474 | 25871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2458 | 2462 | 2461 | 2467 | 9848
  >=65 years | 4005 | 4002 | 4009 | 4007 | 16023
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.1) | 67.1 (7.0) | 67.2 (7.1) | 67.1 (7.1) | 67.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3276 | 3271 | 3271 | 3267 | 13085
  Male | 3187 | 3193 | 3199 | 3207 | 12786
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Not all participants reported race/ethnicity.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 6329 | 6318 | 6324 | 6333 | 25304
    Race/Ethnicity: Non-Hispanic White | 4515 | 4498 | 4529 | 4504 | 18046
    Race/Ethnicity: African-American | 1278 | 1275 | 1271 | 1282 | 5106
    Race/Ethnicity: Hispanic (Not African-American) | 246 | 270 | 245 | 252 | 1013
    Race/Ethnicity: Asian/Pacific Islander | 102 | 86 | 98 | 102 | 388
    Race/Ethnicity: Native American/Alaskan Native | 62 | 56 | 58 | 52 | 228
    Race/Ethnicity: Other/Unknown | 126 | 133 | 123 | 141 | 523
Region of Enrollment [Number; unit: participants]
  United States | 6463 | 6464 | 6470 | 6474 | 25871

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an AMD Event
Description: AMD Event = a composite endpoint of incident AMD plus cases of progression to advanced AMD among participants with AMD at baseline
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin D: Vitamin D3, one 2000 IU capsule/day
- Vitamin D Placebo: Vitamin D placebo, one capsule/day
- Active Omega-3 Fatty Acids: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Omega-3 Fatty Acids Placebo: Omega-3 fatty acids placebo, one capsule/day
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 163 | 161 | 157 | 167
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.82 to 1.27]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.17]

2. Secondary Outcome: Number of Participants With Incident Visually-Significant AMD
Description: AMD responsible for a reduction in best-corrected visual acuity to 20/30 or worse
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 73 | 61 | 61 | 73
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.86 to 1.70]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.59 to 1.17]

3. Secondary Outcome: Number of Participants With Incident Advanced AMD
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 51 | 42 | 39 | 54
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.81 to 1.84]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.48 to 1.09]

4. Other Pre Specified Outcome: Number of Participants With Incident AMD
Description: Incident AMD with or without vision loss to 20/30 or worse; a component of the composite end point of AMD Events
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 148 | 137 | 137 | 148
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.86 to 1.37]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.17]

5. Other Pre Specified Outcome: Number of Participants With AMD Progression
Description: Progression to advanced AMD among participants with AMD at baseline; a component of the composite end point of AMD Events
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 15 | 24 | 20 | 19
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.33 to 1.21]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.56 to 1.97]

6. Other Pre Specified Outcome: Number of Participants With an AMD Event, Excluding the First Two Years of Follow-up
Description: as for outcome 1
Time Frame: 5 years (excluding the first two years of follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 84 | 91 | 83 | 92
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.69 to 1.25]
Statistical Analysis 2: Comparison: Active Omega-3 Fatty Acids vs Omega-3 Fatty Acids Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.67 to 1.21]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Vit D Monitored safety cond'ns: hypercalcemia, kidney stones, parathyroid disease, kidney failure or dialysis; Other symptoms, side effects: GI bleeding, easy bruising; stomach upset or pain; nausea; constipation, diarrhea, skin rash.
  Omega-3 FA Monitored safety cond'ns: GI bleeding; blood in urine; easy bruising; freq nosebleeds; kidney failure or dialysis; Other symptoms, side effects: stomach upset or pain; nausea; constipation; diarrhea; skin rash; bad taste in mouth; increased burping.
Groups:
- Active Vitamin D/Active Omega-3 Fatty Acids: Vitamin D3 (one 2000 IU capsule/day) + Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Active Vitamin D/Placebo Omega-3 Fatty Acids: Vitamin D3, one 2000 IU capsule/day + Omega-3 fatty acids placebo, one capsule/day
- Placebo Vitamin D/Active Omega-3 Fatty Acids: Vitamin D placebo, one capsule/day + Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Placebo Vitamin D/Placebo Omega-3 Fatty Acids: Vitamin D placebo, one capsule/day + Omega-3 fatty acids placebo, one capsule/day
Arm/Group | Active Vitamin D/Active Omega-3 Fatty Acids | Active Vitamin D/Placebo Omega-3 Fatty Acids | Placebo Vitamin D/Active Omega-3 Fatty Acids | Placebo Vitamin D/Placebo Omega-3 Fatty Acids
All-Cause Mortality (participants affected / at risk) | 241/6463 | 244/6464 | 252/6470 | 241/6474
Serious Adverse Events (participants affected / at risk) | 791/6463 | 782/6464 | 822/6470 | 837/6474
Other Adverse Events (participants affected / at risk) | 5101/6463 | 5027/6464 | 5037/6470 | 5101/6474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Active Vitamin D/Active Omega-3 Fatty Acids (N=6463) | Active Vitamin D/Placebo Omega-3 Fatty Acids (N=6464) | Placebo Vitamin D/Active Omega-3 Fatty Acids (N=6470) | Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=6474)
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 170 (170) | 171 (171) | 200 (200) | 203 (203)
Hypercalcemia (Endocrine disorders) | 77 (77) | 70 (70) | 74 (74) | 69 (69)
Invasive cancer of any type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 408 (408) | 385 (385) | 412 (412) | 412 (412) — Total cancer=invasive cancer of any type
Death from cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 75 (75) | 79 (79) | 93 (93) | 94 (94)
Breast cancer (in women) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 60/3276 (60) | 64/3271 (64) | 57/3271 (57) | 65/3267 (65)
Prostate cancer (in men) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 100/3187 (100) | 83/3193 (83) | 110/3199 (110) | 109/3207 (109)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (28) | 23 (23) | 26 (26) | 21 (21)
Major cardiovascular event (Vascular disorders) | 186 (186) | 210 (210) | 200 (200) | 209 (209) — Major cardiovascular event = a composite endpoint of myocardial infarction, stroke, and death from cardiovascular causes
Myocardial infarction (Vascular disorders) | 72 (72) | 97 (97) | 73 (73) | 103 (103)
Stroke (Vascular disorders) | 66 (66) | 75 (75) | 82 (82) | 67 (67)
Death from cardiovascular causes (Vascular disorders) | 74 (74) | 78 (78) | 68 (68) | 70 (70)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Vitamin D/Active Omega-3 Fatty Acids (N=6463) | Active Vitamin D/Placebo Omega-3 Fatty Acids (N=6464) | Placebo Vitamin D/Active Omega-3 Fatty Acids (N=6470) | Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=6474)
Easy bruising (Blood and lymphatic system disorders) | 1737 (1737) | 1697 (1697) | 1706 (1706) | 1702 (1702)
Frequent nosebleeds (Blood and lymphatic system disorders) | 224 (224) | 242 (242) | 241 (241) | 249 (249)
Blood in urine (Blood and lymphatic system disorders) | 469 (469) | 442 (442) | 450 (450) | 432 (432)
Parathyroid condition (Endocrine disorders) | 24 (24) | 26 (26) | 28 (28) | 34 (34) — Parathyroid condition = hyperparathyroidism or hypoparathyroidism
Stomach upset or pain (Gastrointestinal disorders) | 2439 (2439) | 2421 (2421) | 2448 (2448) | 2422 (2422)
Nausea (Gastrointestinal disorders) | 1748 (1748) | 1771 (1771) | 1810 (1810) | 1779 (1779)
Constipation (Gastrointestinal disorders) | 2567 (2567) | 2566 (2566) | 2617 (2617) | 2545 (2545)
Diarrhea (Gastrointestinal disorders) | 2781 (2781) | 2730 (2730) | 2818 (2818) | 2850 (2850)
Increased burping (Gastrointestinal disorders) | 1107 (1107) | 1061 (1061) | 1110 (1110) | 1097 (1097)
Bad taste in mouth (General disorders) | 1109 (1109) | 1086 (1086) | 1131 (1131) | 1159 (1159)
Kidney stones (Renal and urinary disorders) | 233 (233) | 244 (244) | 197 (197) | 229 (229)
Kidney failure or dialysis (Renal and urinary disorders) | 42 (42) | 43 (43) | 43 (43) | 45 (45)
Skin rash (Skin and subcutaneous tissue disorders) | 1629 (1629) | 1639 (1639) | 1702 (1702) | 1728 (1728)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT01782352/Prot_SAP_000.pdf